CLINICAL TRIAL: NCT03094624
Title: Auditory Perceptual and Memory Deficits in Congenital Amusia: Studies of Cerebral Correlates With MEG, Anatomical MRI and Functional MRI
Brief Title: Auditory Deficits in Congenital Amusia (AMUSIE CONGENITALE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0662
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Amusia, Congenital
Keywords: Amusia; Audition; Short-term memory; Emotions; EEG; MEG; MRI
MeSH Terms: conditions — Tune Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amusia (Experimental): Since 2006, recruitment of amusia participants has been organized in the Lyon region, and some 20 participants (and their matched controls in terms of age, sex, laterality, musical practice, number of years of study) have already taken part various studies conducted at the CRNL. The recruitment of amusia participants and controls is continued in order to maintain a sufficient number of participants and compensate for the withdrawals within the cohort already constituted (lack of availability, geographical distance, etc.).
  Interventions: Other: Neuropsychological and neurophysiological tests; Other: Experiment 1; Other: Experiment 2; Other: Experiment 3; Other: Experiment 4
- Matched controls (Sham Comparator): Matched controls of age, sex, laterality, musical practice, number of years of studies.
  Interventions: Other: Neuropsychological and neurophysiological tests; Other: Experiment 1; Other: Experiment 2; Other: Experiment 3; Other: Experiment 4

INTERVENTIONS:
Other: Neuropsychological and neurophysiological tests — Neuropsychological tests consist in listening to sounds in various contexts and providing behavioral responses with response-buttons. Neurophysiological tests consist in the recording of EEG and/or MEG signals or MRI images while realizing the neuropsychological tests, as well as anatomical MRI scanning to characterize the participants' brain anatomy and reconstruct the brain sources of surface EEG/MEG signals.
Other: Experiment 1 — Experiment 1 are interested in perception and musical memory vs. Language and contribute to our understanding of the functional and structural organization of the brain to perceive and memorize music and language.
Other: Experiment 2 — Experiment 2 focuses on perception and musical memory vs. Language and contribute to our understanding of the functional and structural organization of the brain to perceive and memorize music and language. The second experiment will also study short-term memory networks for musical and verbal materials, but the specificity will be the inclusion of a verbal material sung, thus representing the combination of both information. Experiment 2 is divided into two sub-parts. Indeed, the investigators will develop the musical and verbal materials during a first experimental part in experiment (experiment 2a) and then apply them in experimentation MEG (experiment 2b). Experiment 2a will allow us to test new equipment in a short term memory task under conditions that are less restrictive for the participants. Then the investigators will apply the optimal material that emerges for the MEG experiment.
Other: Experiment 3 — Experiment 3 will use Discordant Negativity (MMN; Mismatch Negativity) protocols in coupled EEG-MEG (experiment 3a) and EEG alone (experiment 3b) to investigate memory traces of sensory information. The MMN is used to probe auditory sensory memory (pre-requisite for short- or long-term storage), and has the advantage of being measured without requiring an active task from the participant.
Other: Experiment 4 — Experiment 4 will study the neural correlates of long-term memory for musical and verbal material with fMRI. The testimonies of the amusicians suggest a deficit of the "musical lexicon" which contrasts with that the musical lexicon elaborated of the non-musician listeners.

SUMMARY:
The project studies auditory deficits in congenital amusia at the behavioral and neurophysiological levels.

The auditory processes investigated are pitch discrimination, short-term memory, sound-induced emotions. To characterize auditory deficits in the amusic population, neuropsychological assessments are combined with neurophysiological markers (Electro-encephalography: EEG, Magneto-encephalography: MEG, Magnetic Resonance Imaging: MRI).

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 70 years' old
* French
* Compatibility IRM / MEG (no metal in the body)
* Motivation to participate effectively in the project
* No neurological or psychiatric history
* No severe hearing loss
* Informed consent to participate in the study
* For Amusic participants: participant diagnosed amusic by the MBEA (Montreal Battery of Evaluation of Amusia)
* For Control participants: matched in age, sex, education, music education, laterality, non-amusic (controlled with the MBEA)

Exclusion Criteria:

* Age below 18 or above 70
* Non-Francophone volunteers.
* MRI scanning not possible: artificial cardiac pacemaker, insulin pump, metallic prosthesis, intra-cerebral clip, claustrophobia
* MEG acquisition not possible: large heads, neurostimulator, metal in the head or the body.
* Pregnant or breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-01-13 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Correct answers to the neuropsychological tests | Day 1
  Percentages of correct responses
Neuropsychological tests reaction times | Day 1
  Neuropsychological tests reaction times
Neurophysiological tests EEG | Day 1
  Event-Related Potentials (EEG)
Neurophysiological tests MEG | Day 1
  Event-Related Fields (MEG)
Neurophysiological tests MRI | Day 1
  MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albouy P, Peretz I, Bermudez P, Zatorre RJ, Tillmann B, Caclin A. Specialized neural dynamics for verbal and tonal memory: fMRI evidence in congenital amusia. Hum Brain Mapp. 2019 Feb 15;40(3):855-867. doi: 10.1002/hbm.24416. Epub 2018 Nov 1. PMID 30381866